CLINICAL TRIAL: NCT07070557
Title: High Neutrophil-to-Lymphocyte Ratio and Platelet-to-Lymphocyte Ratio Are Associated With Poor Survival in Patients With Hemodialysis
Brief Title: High Neutrophil-to-Lymphocyte Ratio and Patients With Hemodialysis
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Bassem Ayman Mohamed, resident in internal medicine department, Sohag University
Other Study IDs: Soh-Med--25-6-10MS
Record Dates: First submitted 2025-07-06; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hemodialysis Patient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: neutrophil lymphocyte ratio and platelet lymphocyte ratio — explore the role of neutrophil-to-lymphocyte ratio ( NLR ) and platelet-to-lymphocyte ratio ( PLR ) in predicting mortality in hemodialysis (HD) patients

SUMMARY:
To explore the role of neutrophil-to-lymphocyte ratio ( NLR ) and platelet-to-lymphocyte ratio ( PLR ) in predicting mortality in hemodialysis (HD) patients.

ELIGIBILITY:
Inclusion Criteria:

* All cases with age ≥ 18 years from both sexes female and male, having end-stage renal disease (ESRD), who have been on hemodialysis for at least three months and divided to 4 groups according to the median of NLR and PLR

Exclusion Criteria:

* • Patients aged < 18 years old.

  * Patient with autoimmune disease.
  * Patient with liver cirrhosis.
  * Patients with immunodeficiency.
  * Patients with malignancy.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients on regular hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 6 months
  The primary outcome measures in the study "High Neutrophil-to-Lymphocyte Ratio and Platelet-to-Lymphocyte Ratio Are Associated with Poor Survival in Patients with Hemodialysis" is :- All-cause mortality, encompassing death from any cause These is the endpoint used to evaluate the prognostic significance of NLR and PLR in hemodialysis patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Hemodialysis Unit, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided